CLINICAL TRIAL: NCT06053762
Title: Assessing the Effectiveness of Peer-Facilitated Versus Self-Navigated Tobacco Cessation Interventions for Youths
Brief Title: Identify the Usefulness of Peer-facilitated Versus Self-navigated Quit Tobacco Program for Youths.
Acronym: CEASE Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morgan State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Payam Sheikhattari, Professor, Morgan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB number: #23/04-0093; 5U54MD013376 (NIH)
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Tobacco Product Use
Keywords: Tobacco cessation program, Community-based participatory research, Peer-facilitated approach, Youth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-facilitated tobacco cessation (Experimental): Peer-facilitated tobacco cessation: Participants will be given the evidence-based N-O-T program curriculum for tobacco cessation classes and provided with virtual materials, information, and resources by their assigned peer facilitators. Virtual tobacco cessation peer motivation sessions will be offered using the digital online platform Zoom, and the peer facilitators will communicate with the participants in between the classes Peer-facilitated tobacco cessation: Participants will be given the evidence-based N-O-T program curriculum for tobacco cessation classes and provided with virtual materials, information, and resources by their assigned peer facilitators. Virtual tobacco cessation peer motivation sessions will be offered using the digital online platform Zoom, and the peer facilitators will communicate with the participants in between the classes.
  Interventions: Behavioral: Peer-facilitated tobacco cessation
- Self-navigated tobacco cessation (Other): Self-navigated tobacco cessation: The participants in the self-navigated group will receive the same ALA N-O-T program curriculum and complete the eight-week sessions, but it will be self-navigated and without peer facilitations. No peer facilitator will be assigned to this group and the participants will complete the curriculum by themselves.
  Interventions: Behavioral: Self-navigated tobacco cessation

INTERVENTIONS:
Behavioral: Peer-facilitated tobacco cessation — Peer-facilitated tobacco cessation: Participants will be given the evidence-based N-O-T program curriculum for tobacco cessation classes and provided with virtual materials, information, and resources by their assigned peer facilitators. Virtual tobacco cessation peer motivation sessions will be offered using the digital online platform Zoom, and the peer facilitators will communicate with the participants in between the classes
  Arms: Peer-facilitated tobacco cessation
Behavioral: Self-navigated tobacco cessation — Self-navigated tobacco cessation: The participants in the self-navigated group will receive the same ALA N-O-T program curriculum and will complete the eight-week sessions, but it will be self-navigated and without peer facilitations. No peer facilitator will be assigned to this group and the participants will complete the curriculum by themselves. Self-navigated tobacco cessation: The participants in the self-navigated group will receive the same ALA N-O-T program curriculum and will complete the eight-week sessions, but it will be self-navigated and without peer facilitations. No peer facilitator will be assigned to this group and the participants will complete the curriculum by themselves.
  Arms: Self-navigated tobacco cessation

SUMMARY:
The proposed study is a randomized clinical trial. The overarching goal of the study is to apply Community Based Participatory Research (CBPR) to reduce tobacco use among youth and young adults (14-21 y/o) in Baltimore City through a mixed-method approach adapted to the needs of youth and young adults. This study has partnered with the American Lung Association's Not On Tobacco (N-O-T) program and aims to deliver tobacco cessation classes. The study will target Baltimore City high schools and colleges, prioritizing facilities in underserved inner-city communities. The proposed research consists of a 2-arm trial where participants from four high schools and two colleges will be randomized to peer-facilitated tobacco cessation classes or self-navigated groups. The trial aims to assess the effectiveness of peer-facilitated tobacco cessation intervention compared to self-navigated tobacco cessation in terms of their success rates (quitting and staying quit). The study's primary hypothesis is that the tobacco cessation rate will be equal to or higher in the peer-facilitated arm than in the self-navigated arms. The secondary hypothesis is that the retention rate will be equal to or higher in the peer-facilitated arm compared to the self-navigated arm.

CEASE Youth tobacco cessation program is an eight-week program based on the American Lung Association's (ALA) Not On Tobacco (N-O-T) program. The ALA's N-OT program is acknowledged as an accessible and effective option for teen tobacco cessation. Participants in the peer-facilitated group will be given the evidence-based N-O-T program curriculum and provided with virtual materials, information, and resources by their assigned peer facilitators. Virtual tobacco cessation peer motivation sessions will be offered using the digital online platform Zoom, and the peer facilitators will communicate with the participants in between the classes. The participants in the self-navigated group will receive the same ALA N-O-T program curriculum and complete the eight-week sessions, but it will be self-navigated and without peer facilitations. No peer facilitator will be assigned to this group, and the participants will complete the curriculum by themselves. They will also receive other available resources, including information about the local tobacco cessation services available.

DETAILED DESCRIPTION:
This study is based on the previous CEASE initiative conducted in Baltimore City using a community-based participatory research approach. The study will use a two-arm randomized clinical trial design. Baltimore City high schools and colleges will be randomly allocated to one of the two arms of the study: 1) the peer-facilitated arm and 2) the self-navigated arm.

A list of all identified high schools and colleges will be developed by the research assistant, including those that were engaged during the previous CEASE phases. Based on the characteristics of these schools and colleges, potential eligible partners will be identified, and contact information for each potential partner/site will be obtained. An outreach and engagement consultant will initiate and maintain contact with potential partners/host sites. Targeted outreach messages and resources will be developed and distributed in the form of study information sheet and flyers via email blasts, social media posts, and tabling at school/college events. Once the outreach and engagement consultant establishes contact, members of the research team might be invited to conduct an information session for the partnering school and colleges.

At the information session, interested schools/colleges will receive targeted communications orienting them to the Morgan CARES Network and information about the new iteration of the CEASE program: CEASE Youth. Following all partners' committed engagement or re-engagement, a Partnership Agreement will be developed with each interested entity. This agreement will specify the nature of the engagement (intervention site, recruitment assistance, dissemination activities, etc.) and points of contact for the partnering organization and the CEASE Youth program. The allocation of the host sites to different study arms will be random and blinded and done in a steering committee meeting to ensure the procedure is objective. Following the orientation of school staff, Peer Ambassadors (other high schools or college students) will be recruited, and an orientation and consent process for the peer ambassadors and their parents will be done.

Information sessions will be offered in the various sites as agreed upon with the partners. The information sessions will be offered to a general audience, including prospective participants at events and/or meetings either in-person or virtually via video conference platforms. An information session presentation will be delivered and will describe an overview of the program, eligibility for participation, and the study procedures. Interested high school students will complete a School Survey, which also includes the study eligibility questions, in-person or virtually, using a web-based survey. Participants who are eligible based on the eligibility screening through the school survey will be invited to be enrolled in the study and will complete a registration/enrollment form. Their information will be listed in the enrollment log. Participant IDs will be assigned to participants once they are enrolled in the study. Informed consent will be obtained before starting the intervention. Participating Youths and Young Adults will be recruited either by Peer Ambassadors (other high school or college students) during the first stage of the project (Pre-trial Assessment) or later through advertisement, word of mouth, and referral from school staff.

The data will be collected using forms built in KoboToolbox and will be exported from KoBoToolbox as an Excel file and will be imported to statistical software Stata for cleaning and analysis. The descriptive univariate analysis will be done to review each variable and summarize demographic information. The result will be presented as mean and standard deviation for continuous variables and percentage for categorical variables. The bivariate analysis will be done to compare quit rates with some potential predictor variables using Chi-square tests of independence for categorical variables (gender, race, education, employment) and Student's T-test for continuous variables (age and Fagerstrom score). The results will be presented as numbers with corresponding proportions for the Chi-square tests and presented as means with standard deviations for the T-tests. Multivariate analysis will be done using regression models to compare study outcomes in two study arms. The study will control for several socio-demographic characteristics and other variables. Sub-group analysis will be conducted based on age, gender, race/ethnicity, and other demographic characteristics to compare the effect of the intervention in these different groups.

An Adverse Event Log will be kept by the program manager for each enrolled participant at each intervention site. The program manager will rank each adverse event that is logged by the level of severity, ranging from Mild to Life-Threatening. The likelihood that an adverse event is or is not related to the intervention will also be reported. The CEASE executive committee will outline the appropriate actions to take in response to the adverse event, and potential actions may include: None, Dose Modification, Medical Intervention, Hospitalization, Intervention Discontinued, or Other. The program manager will track and report actions taken. In addition to reporting the outcome of the adverse event, the program manager will also indicate whether or not the event was expected. Adverse events that are reported to be "Severe" or "Life-Threatening" are designated as a "Serious Adverse Event" on the Adverse Event Log as well. Should a Serious Adverse Event (SAE) occur, the program manager will immediately notify the PI. Upon being notified, the PI will complete the Serious Adverse Event Report form detailing the nature of the event and actions taken. All SAEs will be reported in accordance with the Morgan State University IRB procedures and the NIH regulatory and reporting mandates.

The program manager will record events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. At each study visit, the investigator will inquire about the occurrence of AE/SAEs since the last visit. Events will be followed for outcome information until resolution or stabilization.

Adherence to the CEASE intervention will be measured by class attendance. Participants will need to attend the sessions provided in order to benefit from the expected effect of the intervention. The facilitators will record weekly attendance at sessions using the attendance sheet. The attendance records will be used in paying incentives for participation. Participants in both the peer-facilitated and self-navigated arms of the program should complete a maximum of 8 weeks of sessions. At the point of data analysis, all participants enrolled, whether they completed the eight sessions or not, will be included in the data. Participants who attend a total of three sessions out of the eight will, however, be regarded as having poor attendance/compliance in the program because they would not have received enough dosing. Participants who miss two consecutive sessions or three non-consecutive sessions, including the last session, will be regarded as being dropped out of the study. However, every attempt will be taken to follow up with all enrolled participants three months after the end of the intervention. Participants we are unable to reach at this point will be considered lost to follow-up.

The study participant's contact information will be securely stored at Morgan State University's Morgan CARES Center for Urban Health Disparities Research & Innovation, and electronically for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by the MSU IRB or NIMHD requirements. Study participant research data (signed informed consent and photo release forms, school surveys, follow-up surveys etc.) which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the MSU Morgan CARES center and electronically. This will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. Participant IDs will be assigned to participants once they are enrolled into the study. The key list linking the IDs with the participants identifying information will be securely maintained electronically, with access by only the PI, program manager, and selected trained research staff. The Peer facilitators will have sub-lists of the key list for their specific sites/groups, which they will carry safely from the site to their residences and keep properly secured at home until they can bring it to the Morgan CARES center. The security and safety features of the digital communication platforms to be used (Zoom) will be implemented to preserve confidentiality. Zoom meeting IDs will be kept private to the groups only. Passwords or waiting rooms will be used to control access. The study data entry and study management systems used by study sites and by Morgan CARES research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and archived at the Prevention Sciences Research Center (PSRC).

ELIGIBILITY:
Inclusion Criteria:

* Current tobacco user (have used any tobacco product over the past 30 days)
* Individuals who are 14- 21 years old
* Individuals who are ready and willing to quit using tobacco
* Individuals who have access to a digital device (e.g., laptop/computer/tablet) with internet access or data

Exclusion Criteria:

* Individuals who have health conditions preventing them from providing consent will be excluded from the study.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 630 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported tobacco cessation | Self-reported tobacco cessation: 3-5 months post-intervention.
  Self-reported smoking status is a reliable, validated, and widely used measure.

SECONDARY OUTCOMES:
Retention rate | Week 8
  Retention will be measured by the number of sessions attended for the peer-facilitated groups and the number of weeks completed from the curriculum assessed through the weekly check-in form.

CONTACTS AND LOCATIONS:
Locations (1):
- Morgan CARES, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] CDCTobaccoFree. Burden of Tobacco Use in the U.S. Centers for Disease Control and Prevention. Published August 8, 2022. Accessed April 9, 2023. https://www.cdc.gov/tobacco/campaign/tips/resources/data/cigarette-smoking-in-united-states.html
- [Background] National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health. The Health Consequences of Smoking-50 Years of Progress: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK179276/ PMID 24455788
- [Background] Park-Lee E, Ren C, Cooper M, Cornelius M, Jamal A, Cullen KA. Tobacco Product Use Among Middle and High School Students - United States, 2022. MMWR Morb Mortal Wkly Rep. 2022 Nov 11;71(45):1429-1435. doi: 10.15585/mmwr.mm7145a1. PMID 36355596
- [Background] Sun R, Mendez D, Warner KE. Trends in Nicotine Product Use Among US Adolescents, 1999-2020. JAMA Netw Open. 2021 Aug 2;4(8):e2118788. doi: 10.1001/jamanetworkopen.2021.18788. PMID 34432013
- [Background] Ford P, Clifford A, Gussy K, Gartner C. A systematic review of peer-support programs for smoking cessation in disadvantaged groups. Int J Environ Res Public Health. 2013 Oct 28;10(11):5507-22. doi: 10.3390/ijerph10115507. PMID 24169412
- [Background] McKay CE, Dickerson F. Peer Supports for Tobacco Cessation for Adults with Serious Mental Illness: A Review of the Literature. J Dual Diagn. 2012;8(2):104-112. doi: 10.1080/15504263.2012.670847. Epub 2012 May 11. PMID 22904697
- [Background] O'Toole TP, Aaron KF, Chin MH, Horowitz C, Tyson F. Community-based participatory research: opportunities, challenges, and the need for a common language. J Gen Intern Med. 2003 Jul;18(7):592-4. doi: 10.1046/j.1525-1497.2003.30416.x. No abstract available. PMID 12848844
- [Background] Wallerstein, Nina, Duran, Bonnie, Oetzel, John G. and Minkler, Meredith. Community-Based Participatory Research for Health: Advancing Social and Health Equity, 3rd Edition | Wiley. Wiley.com. Accessed April 9, 2023. https://www.wiley.com/en-us/Community+Based+Participatory+Research+for+Health%3A+Advancing+Social+and+Health+Equity%2C+3rd+Edition-p-9781119258858
- [Background] Prado GF, Lombardi EM, Bussacos MA, Arrabal-Fernandes FL, Terra-Filho M, Santos Ude P. A real-life study of the effectiveness of different pharmacological approaches to the treatment of smoking cessation: re-discussing the predictors of success. Clinics (Sao Paulo). 2011;66(1):65-71. doi: 10.1590/s1807-59322011000100012. PMID 21437438
- [Background] Jain A. Treating nicotine addiction. BMJ. 2003 Dec 13;327(7428):1394-5. doi: 10.1136/bmj.327.7428.1394. No abstract available. PMID 14670889
- [Background] Raw M, McNeill A, West R. Smoking cessation: evidence based recommendations for the healthcare system. BMJ. 1999 Jan 16;318(7177):182-5. doi: 10.1136/bmj.318.7177.182. No abstract available. PMID 9888919
- [Background] CDCTobaccoFree. About the Office on Smoking and Health. Centers for Disease Control and Prevention. Published December 2, 2021. Accessed April 9, 2023. https://www.cdc.gov/tobacco/about/osh/index.htm
- [Background] Ramo DE, Liu H, Prochaska JJ. A mixed-methods study of young adults' receptivity to using Facebook for smoking cessation: if you build it, will they come? Am J Health Promot. 2015 Mar-Apr;29(4):e126-35. doi: 10.4278/ajhp.130326-QUAL-128. Epub 2014 Feb 27. PMID 24575728
- [Background] Ranney L, Melvin C, Lux L, McClain E, Lohr KN. Systematic review: smoking cessation intervention strategies for adults and adults in special populations. Ann Intern Med. 2006 Dec 5;145(11):845-56. doi: 10.7326/0003-4819-145-11-200612050-00142. Epub 2006 Sep 5. PMID 16954352
- [Background] Elfeddali I, Bolman C, Candel MJ, Wiers RW, De Vries H. The role of self-efficacy, recovery self-efficacy, and preparatory planning in predicting short-term smoking relapse. Br J Health Psychol. 2012 Feb;17(1):185-201. doi: 10.1111/j.2044-8287.2011.02032.x. Epub 2011 Jun 27. PMID 22107073
- [Background] Bandura A. Social cognitive theory: an agentic perspective. Annu Rev Psychol. 2001;52:1-26. doi: 10.1146/annurev.psych.52.1.1. PMID 11148297
- [Background] Wang TW, Gentzke A, Sharapova S, Cullen KA, Ambrose BK, Jamal A. Tobacco Product Use Among Middle and High School Students - United States, 2011-2017. MMWR Morb Mortal Wkly Rep. 2018 Jun 8;67(22):629-633. doi: 10.15585/mmwr.mm6722a3. PMID 29879097
- [Background] Centers for Disease Control and Prevention (CDC). Tobacco product use among middle and high school students--United States, 2011 and 2012. MMWR Morb Mortal Wkly Rep. 2013 Nov 15;62(45):893-7. PMID 24226625
- [Background] Corey CG, Ambrose BK, Apelberg BJ, King BA. Flavored Tobacco Product Use Among Middle and High School Students--United States, 2014. MMWR Morb Mortal Wkly Rep. 2015 Oct 2;64(38):1066-70. doi: 10.15585/mmwr.mm6438a2. PMID 26421418
- [Background] CDCTobaccoFree. Youth and Tobacco Use. Centers for Disease Control and Prevention. Published November 9, 2022. Accessed April 9, 2023. https://www.cdc.gov/tobacco/data_statistics/fact_sheets/youth_data/tobacco_use/index.htm
- [Background] Wagner FA, Sheikhattari P, Buccheri J, Gunning M, Bleich L, Schutzman C. A Community-Based Participatory Research on Smoking Cessation Intervention for Urban Communities. J Health Care Poor Underserved. 2016;27(1):35-50. doi: 10.1353/hpu.2016.0017. PMID 27763459
- [Background] Sheikhattari P, Zhu S, Clubb PA. New Insights on Tobacco Smoking among the Underserved and Poor. World Academy of Science, Engineering, and Technology. Published online January 1, 2010.
- [Background] Sheikhattari P, Apata J, Kamangar F, Schutzman C, O'Keefe A, Buccheri J, Wagner FA. Examining Smoking Cessation in a Community-Based Versus Clinic-Based Intervention Using Community-Based Participatory Research. J Community Health. 2016 Dec;41(6):1146-1152. doi: 10.1007/s10900-016-0264-9. PMID 27688221
- [Background] Estreet A, Apata J, Kamangar F, Schutzman C, Buccheri J, O'Keefe AM, Wagner F, Sheikhattari P. Improving Participants' Retention in a Smoking Cessation Intervention Using a Community-based Participatory Research Approach. Int J Prev Med. 2017 Dec 19;8:106. doi: 10.4103/ijpvm.IJPVM_303_17. eCollection 2017. PMID 29416835
- [Background] Human Subjects Research Ethics Field Training Guide | Johns Hopkins | Bloomberg School of Public Health. Accessed April 9, 2023. https://publichealth.jhu.edu/offices-and-services/institutional-review-board-irb/training/human-subjects-research-ethics-field-training-guide
- [Background] Cheung KL, de Ruijter D, Hiligsmann M, Elfeddali I, Hoving C, Evers SMAA, de Vries H. Exploring consensus on how to measure smoking cessation. A Delphi study. BMC Public Health. 2017 Nov 21;17(1):890. doi: 10.1186/s12889-017-4902-7. PMID 29162043
- [Background] Moberg J, Kramer M. A brief history of the cluster randomised trial design. J R Soc Med. 2015 May;108(5):192-8. doi: 10.1177/0141076815582303. No abstract available. PMID 26022551
- [Background] Prokhorov AV, Khalil GE, Foster DW, Marani SK, Guindani M, Espada JP, Gonzalvez MT, Idrisov B, Galimov A, Arora M, Tewari A, Isralowitz R, Lapvongwatana P, Chansatitporn N, Chen X, Zheng H, Sussman S. Testing the nicotine dependence measure mFTQ for adolescent smokers: A multinational investigation. Am J Addict. 2017 Oct;26(7):689-696. doi: 10.1111/ajad.12583. Epub 2017 Jul 14. PMID 28708935